CLINICAL TRIAL: NCT07073638
Title: A Phase 2 Trial to Evaluate the Safety and Tolerability and Early Bactericidal Activity of Nebulised RESP30TB in Adults With Newly Diagnosed, Rifampicin Susceptible Pulmonary Tuberculosis
Brief Title: Phase 2 Trial to Evaluate the Safety and Tolerability and Early Bactericidal Activity of RESP30TB in Tuberculosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Thirty Respiratory Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RESP30TB-EBA
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Tuberculoses
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Rifampin; Isoniazid; Pyrazinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RESP30TB (Experimental): Stage 1 - Inhaled RESP30TB 6ml via nebulisation three times daily
  Interventions: Drug: RESP30TB
- RESP30TB + HRZE (Experimental): Stage 2 - Inhaled RESP30TB 6 ml dosed via nebulisation administered three times daily in combination with HRZE taken orally once daily
  Interventions: Drug: RESP30TB; Drug: HRZE (Rifampicin, Isoniazid, Pyrazinamide, Ethambutol combination)

INTERVENTIONS:
Drug: RESP30TB — Nitric Oxide agent
Drug: HRZE (Rifampicin, Isoniazid, Pyrazinamide, Ethambutol combination) — isoniazid 75 mg (H), rifampicin 150 mg (R), pyrazinamide 400 mg (Z), ethambutol 275 mg (E)
  Arms: RESP30TB + HRZE

SUMMARY:
A Phase 2 Trial to Evaluate the Safety and Tolerability and Early Bactericidal Activity of Nebulised RESP30TB in Adults with Newly Diagnosed, Rifampicin Susceptible Pulmonary Tuberculosis

DETAILED DESCRIPTION:
This is a single-centre, open-label, single arm, clinical trial in two sequential stages, with no stratification. 12 patients will be enrolled in Stage 1, and a further 12 patients will be enrolled in Stage 2 (total of 24 patients in the trial).

ELIGIBILITY:
Inclusion Criteria:

1. Provide written, informed consent prior to all trial-related procedures and agree to undergo all trial procedures.
2. Body weight (in light clothing and with no shoes) between 40 and 90 kg, inclusive.
3. Newly diagnosed pulmonary TB.
4. Rifampicin susceptible pulmonary TB as determined by molecular testing.
5. Ability to produce an adequate volume of sputum as estimated from a pre-treatment overnight sputum collection sample (estimated 10 mL or more).
6. Spirometry performed during screening with a Forced Expiration Volume in the first second (FEV1) of ≥ 40%.
7. Be of non-childbearing potential or willing to use effective methods of contraception, as defined in section 4.3.4.

Exclusion Criteria:

1. HIV positive AND CD4 < 350 cells/mm3 OR are receiving antiviral therapy (ART)
2. Baseline Methaemoglobin saturation (SpMet) >3%.
3. Female patients who is pregnant or breast-feeding.
4. Patients planning to conceive a child within the anticipated period of trial participation and for at least 90 days after the last dose of IMP in the trial.
5. Participation in other clinical studies with investigational agents within 8 weeks prior to screening.
6. Treatment received for this episode of TB with any drug active against M.tb
7. Treatment with immunosuppressive medications such as TNF-alpha inhibitors within 2 weeks prior to screening, or systemic corticosteroids for more than 7 days within 2 weeks prior to screening.
8. Treatment with NO and other NO donor agents, phosphodiesterase inhibitors and lung surfactant drugs, within 30 days prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of Inhaled RESP30TB Measured as Number of Treatment Emergent Adverse Events (TEAEs) | Dosing period 14 days + Follow-up period 14 days
  Incidence of Treatment Emergent Adverse Events (TEAEs) will be presented by severity, drug relatedness, seriousness, leading to early withdrawal and leading to death

CONTACTS AND LOCATIONS:
Locations (1):
- TASK Clinical Research Centre, Cape Town, Bellville, South Africa

IPD SHARING:
Plan to Share IPD: No
IPD is confidential until the CSR is published